CLINICAL TRIAL: NCT00001075
Title: A Pilot Study to Evaluate the Immunologic Consequences of a Highly Active Antiretroviral Therapy Regimen (HAART) Consisting of Ritonavir (ABT-538), Zidovudine (AZT), and Lamivudine (3TC) in Moderately Advanced HIV-1 Disease
Brief Title: The Effectiveness of Ritonavir Plus Zidovudine Plus Lamivudine in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 315; 10688 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine; HIV Protease Inhibitors; Ritonavir; Lamivudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Ritonavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Ritonavir
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To determine whether administration of a highly active antiretroviral treatment regimen consisting of ritonavir (ABT-538), zidovudine (AZT), and lamivudine (3TC) is associated with the restoration of delayed type hypersensitivity and lymphocyte proliferative responses in patients with moderately advanced HIV-1 infection. To better characterize in these patients the phenotype of the expanded lymphocyte subpopulations, as well as the genotype, phenotype, and cellular origin of viruses that persist after initiation of therapy, and the genotype and phenotype of drug-resistant isolates that emerge during therapy.

Although plasma viral load drops dramatically after initiation of powerful antiretrovirals, it does not drop to zero. It appears that a new steady state is reached, suggesting that a reservoir may exist of virus-producing cells, possibly cells of monocyte/macrophage lineage, that continue to produce a low level of virus despite antiretroviral treatment.

DETAILED DESCRIPTION:
Although plasma viral load drops dramatically after initiation of powerful antiretrovirals, it does not drop to zero. It appears that a new steady state is reached, suggesting that a reservoir may exist of virus-producing cells, possibly cells of monocyte/macrophage lineage, that continue to produce a low level of virus despite antiretroviral treatment.

Patients undergo 5 weeks of antiretroviral washout before initiating therapy with ritonavir alone for 9 days, followed by combination therapy with ritonavir, zidovudine, and lamivudine from day 10 through week 48. [AS PER AMENDMENT 1/31/97: The availability of the current, open-label study treatment has been extended to allow patients who have completed 48 weeks of therapy to continue protocol therapy until the last enrolled patient completes 48 weeks of study treatment.]

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Recombinant erythropoietin and/or G-CSF for AZT-related bone marrow suppression.
* Antibiotics other than metronidazole.
* PCP prophylaxis.
* Regularly prescribed medications such as antipyretics, analgesics, allergy medicine, and oral contraceptives.
* Vitamins and herbal therapies.

Concurrent Treatment:

Allowed:

* Acupuncture.
* Visualization techniques.

Patients must have:

* Documented HIV infection.
* CD4 count 100-300 cells/mm3.
* At least 3 consecutive months of prior AZT at a dosage of 500-600 mg bid, but with 5 weeks of antiretroviral washout prior to study entry.
* Consent of parent or guardian if less than 18 years old.

Prior Medication:

Required:

* Prior AZT at 500-600 mg bid at any time.
* PCP prophylaxis during antiretroviral washout.

Allowed:

* Prior ddI and/or ddC.
* Prior recombinant erythropoietin and/or G-CSF for AZT-related bone marrow suppression.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Chronic pancreatitis.
* Psychological conditions that would affect compliance.
* Intolerance to 500-600 mg/day AZT.
* Concurrent participation on another antiretroviral research treatment study (study treatment for opportunistic infection or complications of HIV is allowed).
* Considered likely to be noncompliant on study.

Concurrent Medication:

Excluded:

* Immunomodulators such as systemic corticosteroids, thalidomide, or cytokines.
* Rifabutin.
* Disulfiram (Antabuse) or other medications with similar effects, including metronidazole.
* Other drugs contraindicated with ritonavir.

[AS PER AMENDMENT 8/27/96: Immunization must be avoided during the antiretroviral washout period.]

Patients with the following prior conditions are excluded:

* Active opportunistic infection or febrile illness with temperature >= 38.5 C within 3 days prior to study entry.
* History of acute pancreatitis within the past 2 years.

Prior Medication:

Excluded:

* Prior 3TC or a protease inhibitor.
* Experimental drugs except those for HIV-related conditions, within the past 30 days.

[AS PER AMENDMENT 8/27/96: Immunization must be avoided prior to the antiretroviral washout period.]

Active substance abuse.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55
Dates: Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lederman M, Study Chair; Kessler H, Study Chair
Locations (3):
- United States (3):
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Case CRS, Cleveland, Ohio

REFERENCES:
- [Background] Connick E, Lederman MM, Kotzin BL, Spritzler J, Kuritzkes DR, St Clair M, Sevin AD, Fox L, Chiozzi MH, Leonard JM, Rousseau F, D'Arc Roe J, Martinez A, Kessler H, Landay A. Immune reconstitution in the first year of potent antiretroviral therapy and its relationship to virologic response. J Infect Dis. 2000 Jan;181(1):358-63. doi: 10.1086/315171. PMID 10608789
- [Background] Lederman MM, Connick E, Landay A, Kuritzkes DR, Spritzler J, St Clair M, Kotzin BL, Fox L, Chiozzi MH, Leonard JM, Rousseau F, Wade M, Roe JD, Martinez A, Kessler H. Immunologic responses associated with 12 weeks of combination antiretroviral therapy consisting of zidovudine, lamivudine, and ritonavir: results of AIDS Clinical Trials Group Protocol 315. J Infect Dis. 1998 Jul;178(1):70-9. doi: 10.1086/515591. PMID 9652425
- [Background] Kaushal S, Landay AL, Lederman MM, Connick E, Spritzler J, Kuritzkes DR, Kessler H, Levine BL, St Louis DC, June CH. Increases in T cell telomere length in HIV infection after antiretroviral combination therapy for HIV-1 infection implicate distinct population dynamics in CD4+ and CD8+ T cells. Clin Immunol. 1999 Jul;92(1):14-24. doi: 10.1006/clim.1999.4726. PMID 10413649
- [Background] Kuritzkes DR, Sevin A, Young B, Bakhtiari M, Wu H, St Clair M, Connick E, Landay A, Spritzler J, Kessler H, Lederman MM. Effect of zidovudine resistance mutations on virologic response to treatment with zidovudine-lamivudine-ritonavir: genotypic analysis of human immunodeficiency virus type 1 isolates from AIDS clinical trials group protocol 315.ACTG Protocol 315 Team. J Infect Dis. 2000 Feb;181(2):491-7. doi: 10.1086/315244. PMID 10669331
- [Background] Doepel L, Folkers G. NIAID researchers present new findings at retrovirus meeting. National Institute of Allergy and Infectious Diseases. NIAID AIDS Agenda. 1997 Mar:4, 11. PMID 11364173
- [Background] Shapiro HM, Lederman M, Connick E, Kessler H, Kuritzkes DR, Landay AL. Small differences in CD4+ T-cell production may go unnoticed. AIDS. 1999 Feb 4;13(2):290-1. doi: 10.1097/00002030-199902040-00025. No abstract available. PMID 10202843
- [Background] ACTG 315 drug cocktail restores immune function. AIDS Patient Care STDS. 1997 Jun;11(3):193. doi: 10.1089/apc.1997.11.193. No abstract available. PMID 11361794
- [Background] Wu H, Connick E, Kuritzkes DR, Landay A, Spritzler J, Zhang B, Spear GT, Kessler H, Lederman MM; ACTG 315 Team. Multiple CD4+ cell kinetic patterns and their relationships with baseline factors and virological responses in HIV type 1 patients receiving highly active antiretroviral therapy. AIDS Res Hum Retroviruses. 2001 Sep 1;17(13):1231-40. doi: 10.1089/088922201750461285. PMID 11559422
- [Background] Lederman M, Connick E, Landay A, Kessler H, Kuritzkes D, St Clair M, Fox L, Heath-Chiozzi M, Rousseau F, Spritzler J. Partial immune reconstitution after 12 weeks of HAART (AZT, 3TC, ritonavir) preliminary results of ACTG 315. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:208 (abstract no LB13)
- [Background] Wu H, Kuritzkes DR, McClernon DR, Kessler H, Connick E, Landay A, Spear G, Heath-Chiozzi M, Rousseau F, Fox L, Spritzler J, Leonard JM, Lederman MM. Characterization of viral dynamics in human immunodeficiency virus type 1-infected patients treated with combination antiretroviral therapy: relationships to host factors, cellular restoration, and virologic end points. J Infect Dis. 1999 Apr;179(4):799-807. doi: 10.1086/314670. PMID 10068574
- [Derived] Gillespie EA, Gillespie BW, Stevens MJ. Painful diabetic neuropathy: impact of an alternative approach. Diabetes Care. 2007 Apr;30(4):999-1001. doi: 10.2337/dc06-1475. No abstract available. PMID 17392561